CLINICAL TRIAL: NCT06152731
Title: HRD Tests for Ovarian cancER
Acronym: HERO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A01585-40
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer
Keywords: HRD (Homologous Recombination Deficient); GIScar; myChoice; platinum chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Kenny-Caffey syndrome, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HRD tests (Other): To determine HRD status on the tumor, 2 different tests will be used concomitantly
  Interventions: Genetic: tests to determine HRD status

INTERVENTIONS:
Genetic: tests to determine HRD status — Test Giscar AND test myChoice will be performed.
  If one or two tests identifies a HRD status :
  a PARP inhibitor treatment may be initiated according to current recommendations

SUMMARY:
The study concerns patients with Invasive epithelial ovarian cancer, primary Fallopian tube carcinoma, ovarian-type peritoneal carcinoma, and with an indication of a first-line platinum-based chemotherapy.

To determine HRD status, 2 separate tests will be performed in the study:

1. Giscar assay : developed by the sponsor
2. myChoice assay

If one or two tests identifies a HRD status :

a PARP inhibitor treatment may be initiated according to current recommendations

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-year or more
* Histologically documented high grade serous epithelial ovarian cancer, fallopian tube or peritoneum cancer
* Newly diagnosed advanced (International Federation of Gynecology and Obstetrics [FIGO] stage III or IV) ovarian carcinoma, candidate to a first line platinum-based chemotherapy
* Tumor tissue must be available for HRD analyses (FFPE tissue block) and

  * Collected if possible during the initial surgery or the initial biopsy (before chemotherapy)
  * With sufficient tumour surface area (> 25 mm²), with a final cellularity of at least 20%
* Patient affiliated to an appropriate social security system
* Patient signed consent form before any trial related activities

Exclusion Criteria:

* Recurrent high grade serous epithelial ovarian cancer, fallopian tube or peritoneum cancer
* Non epithelial or borderline ovarian cancer
* Other tumor, for which the treatment may interfere with the ovarian cancer treatment and/or that may have a major impact on prognosis
* Exclusive palliative setting
* Patient deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Rate of platinum-sensitive ovarian cancer patients according to GIScar HRD signature (classified into HRD or HRP). | six months after the end of platinum-based chemotherapy
  Evaluate Platinum-sensitivity patients (defined as absence of disease progression, according to RECIST 1.1 criteria, six months after a first-line platinum-based chemotherapy) correlated with Homologous Recombination status in tumor (HRD : Homologous Recombination deficient / HRP :Homologous Recombination Proficient)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Chu Amiens, Amiens
  - Centre Francois Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leman R, Cherifi F, Leheurteur M, Theret P, Pasquesoone C, Saint-Ghislain M, Bresson L, Denoyelle C, Vigneron N, Poulain L, Delepee R, Berby B, Dremaux J, Dumont A, Blanc-Fournier C, Jeanne C, Briand M, Rousseau N, Pepin LF, Deruche E, Dumont F, Leconte A, Lequesne J, Clarisse B, Joly F, Castera L, Rouzier R. Homologous recombination deficiency (HRD) tests for ovarian cancer: a multicenter French phase II study (HERO). BMC Cancer. 2025 Jul 1;25(1):1075. doi: 10.1186/s12885-025-14423-2. PMID 40597907